CLINICAL TRIAL: NCT04338282
Title: Maintenance Therapy With Anti-PD-1 Antibody for Patients With NK/T-cell Lymphoma: a Single Arm, Single Center, Open Label, Phase 2 Trial
Brief Title: Maintenance Therapy With Anti-PD-1 Antibody for Patients With NK/T-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, LIANG WANG, Director of department of hematology, Beijing Tongren Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRhos-ENKTCL-5
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Extranodal NK/T-cell Lymphoma, Nasal Type
Keywords: extranodal NK/T-cell lymphoma; PD-1 blockade; maintenance therapy
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — toripalimab; spartalizumab

STUDY DESIGN:
Intervention Model Description: For patients with positive plasma EBV-DNA at the end of treatments, anti-PD-1 antibody (toripalimab 240mg, every 3 weeks for up to one year)is given as maintenance therapy for 1 year.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): anti-PD-1 antibody (toripalimab) 240mg/d, every 3 weeks, for up to one year or until disease progression.
  Interventions: Drug: toripalimab

INTERVENTIONS:
Drug: toripalimab — 240mg/d, every 3 weeks, for up to one year or until disease progression, whichever comes first
  Other Names: anti-PD-1-antibody

SUMMARY:
For patients with NK/T-cell lymphoma, plasma EBV-DNA has been found to be a prognostic factor, and those with positive plasma EBV-DNA at the end of treatments are more likely to suffer from disease relapse. Thus, this study aims to evaluate the role of maintenance with anti-PD-1 antibody.

DETAILED DESCRIPTION:
For patients with NK/T-cell lymphoma, plasma EBV-DNA has been found to be a prognostic factor, and those with positive plasma EBV-DNA at the end of treatments are more likely to suffer from disease relapse. The investigators previously reported one-year progression free survival rate of 22.2% for patients with positive plasma EBV-DNA at the end of treatments. Recently, anti-PD-1 antibody has been shown to be highly effective in the treatment of NK/T-cell lymphoma. Thus, this study aims to evaluate the role of maintenance with anti-PD-1 antibody for patients with positive plasma EBV-DNA at the end of treatments.

ELIGIBILITY:
Inclusion Criteria:

* Pathology confirmed diagnosis of NK/T-cell lymphoma.
* Plasma EBV-DNA was positive at the end of first-line pegaspargase-based regimens.
* ECOG score of 0-3 points.
* The lab tests within 1 week before enrollment meets the following:

  * Blood routine: Hb≥80g/L, PLT≥50×10e9/L.
  * Liver function: ALT, AST, TBIL≤2 times the upper limit of normal.
  * Renal function: Cr is normal.
  * Coagulation: plasma fibrinogen≥1.0g/L.
  * Cardiac function: LVEF≥50%, ECG is normal
* Sign the informed consent form.
* Voluntary compliance with research protocols.

Exclusion Criteria:

* Patients had relapsed NK/T-cell lymphoma.
* Active infection requires ICU treatment.
* Concomitant HIV infection or active infection with HBV, HCV.
* Serious complications such as fulminant DIC.
* Significant organ dysfunction:

  * respiratory failure
  * NYHA classification≥2 chronic congestive heart failure
  * decompensation Hepatic or renal insufficiency
  * high blood pressure and diabetes that cannot be controlled
  * cerebral vascular events within the past 6 months.
* Pregnant and lactating women.
* Had a history of autoimmune diseases, and disease was active now. Those who were known to be allergic to drugs in the study regimen.
* Patients with other tumors who require treatments within 6 months.
* Other experimental drugs are being used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
one-year progression free survival rate | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  progression free survival is caculated from date of study enrollment to documented disease progression or death of any reason, whichever came first

SECONDARY OUTCOMES:
one-year overall survival rate | From date of enrollment until the date of documented death from any cause or last follow up, whichever came first, assessed up to 12 months
  overall survival is caculated from date of study enrollment to documented death of any reason or last follow up, whichever came first
negative conversion rate of plasma EBV-DNA | up to one year
  plasma EBV-DNA status converted from positive to negative

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wang L, Wang H, Wang JH, Xia ZJ, Lu Y, Huang HQ, Jiang WQ, Zhang YJ. Post-treatment plasma EBV-DNA positivity predicts early relapse and poor prognosis for patients with extranodal NK/T cell lymphoma in the era of asparaginase. Oncotarget. 2015 Oct 6;6(30):30317-26. doi: 10.18632/oncotarget.4505. PMID 26210287